CLINICAL TRIAL: NCT03172429
Title: Cerebral Tissue Oxygenation in Highlanders With Pulmonary Hypertension Compared to Highlanders Without Pulmonary Hypertension and Lowlanders
Brief Title: Cerebral Tissue Oxygenation in Highlanders/Lowlanders
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: National Center of Cardiology and Internal Medicine named after academician M.Mirrakhimov (Other Government)
Responsible Party: Sponsor
Other Study IDs: 01-8/433C
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: High Altitude Pulmonary Hypertension
Keywords: pulmonary hypertension; cerebral tissue oxygenation; disease progression; hypoxia
MeSH Terms: conditions — Pulmonary edema of mountaineers; Hypertension, Pulmonary; Disease Progression; Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- High altitude pulmonary hypertension: Highlanders with high altitude pulmonary hypertension living above 2500 m.
- High altitude control: Healthy highlanders living above 2500 m.
- Low altitude control: Healthy lowlanders living below 1000 m.

SUMMARY:
The purpose of the current study is to evaluate the cerebral tissue oxygenation of Kyrgyz highlanders with high altitude pulmonary hypertension (HAPH) by performing a longitudinal cohort study. To this end, the investigators will invite the same highlanders who participated in the study in 2012 to undergo follow-up examinations in 2017, in order to allow comparisons of current results with baseline data from 2012.

ELIGIBILITY:
Inclusion Criteria:

* high altitude pulmonary hypertension confirmed by clinical presentation and mean pulmonary artery pressure >30 mmHg measured by echocardiography at altitude of residence.
* healthy subjects (high altitude controls)
* Both genders
* Age >16 y
* Kyrgyz ethnicity
* born, raised and currently living at >2500 m
* healthy subjects currently living at <1000 m (low altitude controls)

Exclusion Criteria:

* Pulmonary hypertension from other causes, in particular from left ventricular failure as judged clinically and by echocardiography
* Excessive erythrocytosis
* Other coexistent disorders that may interfere with the cardio-respiratory system and sleep
* Regular use of medication that affects control of breathing
* Heavy smoking

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Highlanders with high altitude pumonary hypertension living at an altitude of 2500-4000 m; healthy highlanders living at an altitude of 2500-4000 m; healthy lowlanders living at an altitude of <1000 m.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-05-24 (Actual); Primary Completion 2017-08-16 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
Changes in cerebral tissue oxygenation | Year 2012 to 2017
  Difference in the change in cerebral tissue oxygenation (CTO, measured by near infrared spectroscopy) 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander

SECONDARY OUTCOMES:
Changes in cerebrovascular response to hyperoxia | Year 2012 to 2017
  Difference in the change in cerebrovascular response (total hemoglobin concentration, a surrogate to blood volume, measured by near infrared spectroscopy) to hyperoxia 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Changes in cerebrovascular response to hypocapnia | Year 2012 to 2017
  Difference in the change in cerebrovascular response (total hemoglobin concentration, a surrogate to blood volume, measured by near infrared spectroscopy) to hypocapnia 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander
Arterial oxygen saturation | Year 2012 to 2017
  Difference in the change in the arterial oxygen saturation 2012 to 2017 in highlanders with high altitude pulmonary hypertension, healthy highlanders and healthy lowlander

CONTACTS AND LOCATIONS:
Overall Officials: Talant M Sooronbaev, MD, Study Chair — NCCIM
Locations (1):
- National Center for Cardiology and Internal Medicine, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided